CLINICAL TRIAL: NCT06103890
Title: A Study on Dynamic Monitoring of ctDNA in Neoadjuvant Therapy With Cetuximab Combined With Albumin-bound Paclitaxel and Nedaplatin for Esophageal Squamous Cell Carcinoma
Brief Title: Dynamic ctDNA Monitoring in Neoadjuvant Therapy for Esophageal Squamous Cell Carcinoma
Acronym: ctDNA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hebei Medical University Fourth Hospital (Other)
Collaborators: Handan Central Hospital (Other); Xingtai People's Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: NATEC
Record Dates: First submitted 2023-09-13; First posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Esophageal Squamous Cell Carcinoma
Keywords: neoadjuvant therapy; esophageal squamous cancer; ctDNA; immunochemotherapy; dynamic monitoring; biomarker
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study is a prospective, multicenter, open-label, observational cohort study. The primary endpoint is pathological complete response (pCR), and the secondary endpoints include R0 resection rate, ctDNA clearance rate, major pathological response (MPR), recurrence-free survival (RFS), and overall survival (OS). Chinese patients with esophageal squamous cell carcinoma who are eligible for surgical resection will receive neoadjuvant therapy with cetuximab combined with albumin-bound paclitaxel and nedaplatin. Personalized ctDNA monitoring will be conducted at multiple time points, including before neoadjuvant therapy, during therapy, preoperatively, postoperatively, and during adjuvant therapy, to explore the clinical value of minimal residual disease (MRD) as a biomarker for assessing treatment efficacy, predicting recurrence risk, and evaluating prognosis in esophageal squamous cell carcinoma. This study aims to enroll 100 Chinese patients with stage II-III (potentially) resectable esophageal squamous cell carcinoma.

DETAILED DESCRIPTION:
This study aims to enroll 100 Chinese patients with stage II-III (potentially) resectable esophageal squamous cell carcinoma.

Tumor tissue samples will be collected from the subjects before neoadjuvant therapy for whole-exome sequencing (WES). Based on the WES results, personalized ctDNA detection panels will be designed (referred to as panel 1) for blood-based multiplex PCR-NGS testing. Blood samples will be collected at baseline (T0), after the first cycle of treatment (T1), after the second cycle of treatment (T2), after the third cycle of treatment (T3), and after the fourth cycle of treatment (T4) for monitoring.

Intraoperative tumor tissue will be collected. For patients with tumor cell content ≥20%, WES will be performed, and a personalized ctDNA detection panel (referred to as panel 2) will be designed based on the WES results. For patients with tumor cell content <20%, panel 1 will continue to be used for blood-based multiplex PCR-NGS testing. Blood samples will be collected before surgery (T5), 3-7 days after surgery (T6), and during the adjuvant therapy period (T7-TN) for ctDNA monitoring. MRD monitoring will be conducted every 3-6 months during follow-up, with dynamic recurrence monitoring until radiological recurrence or the end of the study. The stable detection limit for ctDNA monitoring is 0.02%.

It is expected to complete enrollment within 1 year. Clinical and pathological data, such as performance status, imaging, and serum markers (e.g., CEA), will be collected during the clinical trial. Follow-up will be conducted for 24 months, and data on treatment regimens, recurrence-free survival (RFS), overall survival (OS), adverse events (AE), etc., will be collected. Continuous observation will be conducted for up to 3 years.

Bioinformatics analysis will be performed on the data to construct mutation profiles. Statistical analysis will be conducted to establish the correlation between ctDNA positivity, mutation characteristics, and prognostic indicators. The ctDNA data analysis results will be linked to clinical management to ultimately improve clinical care.

Treatment regimen: Neoadjuvant therapy with cetuximab combined with albumin-bound paclitaxel and nedaplatin for 2-4 cycles:

Albumin-bound paclitaxel: 400mg, IV, on day 1, every 3 weeks; Nedaplatin: 80 mg/m2, IV, every 3 weeks; Cetuximab: 200mg, IV, on day 1, every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 and 70 years, regardless of gender.
2. Patients with histologically confirmed clinical stage II-III thoracic esophageal squamous cell carcinoma.
3. Neck enhanced CT scan showing no suspicious lymph node metastasis in the neck; no systemic metastasis detected by imaging examination.
4. Expected to achieve R0 resection.
5. ECOG performance status of 0-1.
6. No prior anti-tumor treatment for esophageal cancer, including chemotherapy, radiotherapy (including planned radiotherapy during the study period), hormone therapy, and immunotherapy.
7. Measurable lesions (according to RECIST v1.1 criteria).
8. Preoperative evaluation of organ function shows no contraindications for surgery.
9. Laboratory tests confirm good bone marrow, liver, kidney function, and coagulation function.
10. Able to provide informed consent and willing to cooperate with clinical follow-up.
11. Willing to provide peripheral blood samples for testing, as well as the patient's medical history, current treatment information, imaging studies, and tumor marker data, and willing to use the testing data for further scientific research, clinical diagnosis and treatment, and commercial product development.

Exclusion Criteria:

1. Unable to provide a sufficient amount of tissue samples/blood samples required for the study before treatment.
2. Patient refuses to undergo MRD testing.
3. History of malignancies other than esophageal cancer within the past 5 years (excluding cured localized tumors, such as cervical carcinoma in situ, basal cell carcinoma, and prostate carcinoma in situ; patients with prostate cancer who have received hormone therapy and achieved disease-free survival for more than 5 years are not excluded).
4. History of gastrointestinal bleeding within the past 6 months, or presence of coagulation abnormalities at enrollment, or currently receiving thrombolytic or anticoagulant therapy, indicating a high risk of bleeding.
5. Severe cardiovascular or cerebrovascular diseases.
6. History of interstitial lung disease or active pneumonia requiring steroid treatment at enrollment.
7. Active tuberculosis at enrollment or received anti-tuberculosis treatment within the past year.
8. Bronchial asthma requiring intermittent use of bronchodilators or other medical interventions at enrollment.
9. Presence of systemic infectious diseases requiring systemic treatment within the past 4 weeks at enrollment.
10. Severe unhealed wounds, active ulcers, or untreated fractures at enrollment.
11. Presence of other non-surgical conditions.
12. Previous surgeries that prevent the use of gastric conduit for esophageal reconstruction.
13. Severe allergic reactions to chemotherapy drugs (such as paclitaxel, albumin-bound paclitaxel, cisplatin, or carboplatin) or any monoclonal antibody.
14. History of organ transplantation.
15. Other conditions deemed unsuitable for participation in this study according to the investigator's judgment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with stage II-III (potentially) operable esophageal squamous cell carcinoma
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-05-22 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
pCR | Up to 1 year
  pCR stands for pathological complete response. It refers to the absence of any detectable cancer cells in the tissue sample taken during surgery after neoadjuvant treatment.

SECONDARY OUTCOMES:
R0 resection rate | Up to 1 year
  The R0 resection rate refers to the rate of complete tumor removal without any residual tumor cells in the surgical specimen after neoadjuvant treatment.
ctDNA clearance rate | Up to 1 year
  The ctDNA clearance rate refers to the extent of elimination of circulating tumor DNA (ctDNA) during neoadjuvant treatment. It is evaluated by comparing the levels of ctDNA before and after neoadjuvant therapy to assess the impact of treatment on the tumor.
MPR | Up to 1 year
  MPR stands for Major Pathological Response. It refers to a significant reduction or disappearance of tumor cells in the surgical specimen after neoadjuvant therapy.
RFS | 3 years
  RFS stands for Recurrence-Free Survival. It refers to the length of time after curative surgery following neoadjuvant treatment during which a patient remains free from any signs or symptoms of cancer recurrence.
OS | 3 years
  OS stands for Overall Survival. It refers to the length of time from the start of neoadjuvant treatment to the death of a patient from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Ziqiang Tian, MD, Study Chair — Department of Thoracic Surgery, Fourth Hospital of Hebei Medical University
Locations (1):
- Department of Thoracic Surgery, Fourth Hospital of Hebei Medical University, Shijiazhuang, Hebei, China